CLINICAL TRIAL: NCT02908191
Title: A Phase 1a/1b, Dose-Ranging Study of the Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of ABI-H0731 in Healthy Volunteers and Patients With Chronic Hepatitis B
Brief Title: A Study in Healthy Volunteers and Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABI-H0731-101
Record Dates: First submitted 2016-09-14; First posted 2016-09-20 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Sugars; entecavir; Tenofovir; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABI-H0731 or Matching Placebo (Experimental): ABI-H0731 in varying doses of tablets by mouth for 1 day, 7 days, or 28 days
  Interventions: Drug: ABI-H0731; Drug: Placebo for ABI-H0731
- ABI-H0731 or Placebo and ETV or TDF (Experimental): ABI-H0731 and entecavir or tenofovir in combination in a yet to be determined dose by mouth for 28 days
  Interventions: Drug: ABI-H0731; Drug: Placebo for ABI-H0731; Drug: Entecavir; Drug: Tenofovir disoproxil fumarate
- ABI-H0731 or Placebo and a Nucleos(t)ide and Pegasys (Experimental): ABI-H0731 or Placebo, in combination with a commerically-approved nucleos(t)ide plus PegIFN in treatment-experienced patients, for 28 days
  Interventions: Drug: ABI-H0731; Drug: Placebo for ABI-H0731; Drug: Pegasys; Drug: Nucleos(t)ide

INTERVENTIONS:
Drug: ABI-H0731
Drug: Placebo for ABI-H0731
  Other Names: Sugar pill manufactured to mimic the ABI-H0731 tablet
Drug: Entecavir — Used to treat adults with chronic hepatitis B virus
  Arms: ABI-H0731 or Placebo and ETV or TDF
Drug: Tenofovir disoproxil fumarate — Used to treat adults with chronic hepatitis B virus
  Arms: ABI-H0731 or Placebo and ETV or TDF
Drug: Pegasys — Used to treat adults with chronic hepatitis B virus who show signs of liver damage
  Other Names: peginterferon alfa-2a
  Arms: ABI-H0731 or Placebo and a Nucleos(t)ide and Pegasys
Drug: Nucleos(t)ide — Used to treat adults with chronic hepatitis B virus
  Arms: ABI-H0731 or Placebo and a Nucleos(t)ide and Pegasys

SUMMARY:
This two-part, Phase 1 protocol will be the first clinical study of ABI-H0731. Part I will be a Phase 1a dose-ranging assessment of ABI-H0731 in healthy adult volunteers. If the dose-related safety, tolerability and pharmacokinetics (PK) of ABI-H0731 in human volunteers are deemed satisfactory, then the study will advance to Part II, a Phase 1b dose-ranging assessment of ABI-H0731 in non-cirrhotic, CHB patients.

ELIGIBILITY:
Healthy volunteers:

1. Male or female between 18 and 65 years old with a BMI of 18-32kg/m2
2. Must be in good health and not have any health condition which could interfere with the absorption, distribution or elimination of study drug, or with the clinical and laboratory assessments in this study

CHB patients:

1. Male or female between 18 and 65 years of age, with a BMI of 18-35kg/m2 and a minimum body weight of 45 kg
2. Must have chronic hepatitis B with no history of clinical decompensation
3. Seropositive for HIV, HCV, or HDV antibody at Screen
4. Previous treatment with any HBV antiviral treatments within the last 3 months
5. Other known cause of liver disease, including NASH

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Number of healthy volunteers and patients with chronic HBV infection with treatment-related adverse events as assessed by CTCAE v4.0. | Up to 57 days

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Auckland
  - Hamilton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yuen MF, Agarwal K, Gane EJ, Schwabe C, Ahn SH, Kim DJ, Lim YS, Cheng W, Sievert W, Visvanathan K, Ruby E, Liaw S, Yan R, Huang Q, Colonno R, Lopatin U. Safety, pharmacokinetics, and antiviral effects of ABI-H0731, a hepatitis B virus core inhibitor: a randomised, placebo-controlled phase 1 trial. Lancet Gastroenterol Hepatol. 2020 Feb;5(2):152-166. doi: 10.1016/S2468-1253(19)30346-2. Epub 2019 Nov 9. PMID 31711752